CLINICAL TRIAL: NCT02665026
Title: A Single Center, Open, Randomized Clinical Trials, Effectiveness and Safety Study on Different Timing of Preventive Ileostomy Closure After Total Mesorectal Excision for Middle and Low Rectal Cancer
Brief Title: Effectiveness and Safety Study on Different Timing of Preventive Ileostomy Closure After Surgery for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jianbin Xiang, professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2015-276
Record Dates: First submitted 2016-01-23; First posted 2016-01-27 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stoma closure at different times (Experimental): choose different times to do stoma closure after surgery for rectal cancer
  Interventions: Procedure: stoma closure at different times

INTERVENTIONS:
Procedure: stoma closure at different times — Early closure: stoma closure in 12 weeks after surgery for rectal cancer; Late group: stoma closure in 24 weeks after surgery for rectal cancer

SUMMARY:
The purpose of this study is to evaluate the appropriate timing to do preventive ileostomy closure after total mesorectal excision of rectal cancer. To evaluate the effectiveness and safety of preventive ileostomy closure at different time (12 weeks / 24 weeks after radical resection of rectal carcinoma). This study was expected to demonstrate that the early preventive ileostomy closure after total mesorectal excision of rectal cancer does not increase the risk of complications.

DETAILED DESCRIPTION:
A temporary stoma may, in fact, result in reduced quality of life because of feelings of physical and mental restriction, debilitating nuisance, among other problems. Skin irritation, prolapse, and retractionare quite common after ileostomy. A high incidence of parastomal hernia, ileus, and increased salt and fluid loss has been reported, which may also contribute to greater willingness of both the surgeon and patient to close the temporary stoma as soon as possible.

Currently, it remains unclear whether stoma closure should be performed after the end of chemotherapy or during chemotherapy (12 weeks or 24 weeks after radical resection of rectal carcinoma).

The aim of this study is to assess the possible impact of stoma closure timing on postoperative results and to evaluate that the early preventive ileostomy closure after total mesorectal excision of rectal cancer does not increase the risk of complications.

ELIGIBILITY:
Inclusion Criteria:

* sign the informed consent
* postoperative pathology is rectal adenocarcinoma
* primary middle and low rectal cancer patients (tumor distance from the anal margin is less than 10 cm)
* underwent total mesorectal excision for rectal cancer with preventive loop ileostomy

Exclusion Criteria:

* postoperative pathology is not rectal adenocarcinoma (rectal neuroendocrine tumor, lymphoma, etc.)
* postoperative pathologic staging of rectal cancer is I phase, II phase
* underwent total mesorectal excision for rectal cancer without preventive loop ileostomy
* emergency operation for rectal cancer
* disease progression (local recurrence or distant metastasis, etc.)
* anastomotic stenosis
* serious system disease, including heart dysfunction, respiratory insufficiency, liver and kidney dysfunction, serious blood diseases
* participate in other clinical trial
* pregnancy or perinatal woman
* combined with other malignant tumor
* with a history of neurological and psychiatric disorders
* patients with abnormal bone marrow suppression after chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complication | within the first 2 weeks after surgery

SECONDARY OUTCOMES:
Postoperative quality of life | five years
survival rate | five years
Disease-free survival | five years

CONTACTS AND LOCATIONS:
Overall Officials: Jianbin Xiang, doctor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for all primary and secondary outcome measures will be made available within 6 months of study completion.

REFERENCES:
- [Background] Matthiessen P, Hallbook O, Rutegard J, Simert G, Sjodahl R. Defunctioning stoma reduces symptomatic anastomotic leakage after low anterior resection of the rectum for cancer: a randomized multicenter trial. Ann Surg. 2007 Aug;246(2):207-14. doi: 10.1097/SLA.0b013e3180603024. PMID 17667498
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Tulchinsky H, Shacham-Shmueli E, Klausner JM, Inbar M, Geva R. Should a loop ileostomy closure in rectal cancer patients be done during or after adjuvant chemotherapy? J Surg Oncol. 2014 Mar;109(3):266-9. doi: 10.1002/jso.23493. Epub 2013 Nov 19. PMID 24249401